CLINICAL TRIAL: NCT01582243
Title: A Prospective, Open-label, Interventional Study to Assess the HbA1c Change an 24-hr Glucose Fluctuation After Vildagliptin Plus Metformain (SPC) Treatment in Metformin Monotherapy Uncontrolled Type 2 Diabetes Mellitus Patients
Brief Title: Safety and Efficacy of Vildagliptin Plus Metformin (SPC) Treatment in Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ATW03
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, type 2; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

ARMS (1):
- Vildagliptin plus metformin (SPC) (Experimental): Eligible participants received oral vildagliptin 50 mg plus metformin 500 mg (SPC) twice daily from week 1 to week 24.
  Interventions: Drug: Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin 50 mg plus metformin 500 mg as Single Pill combination (SPC)
  Other Names: LAF237, Galvus Met

SUMMARY:
This study will assess the efficacy of vildagliptin plus metformin (SPC) treatment in type 2 diabetes mellitus patients uncontrolled by metformin monotherapy after 24 weeks treatment

ELIGIBILITY:
Inclusion criteria

1. Outpatients who were 20 years of age and older with diagnosis of T2DM.
2. Patients who had been treated with stable dose of metformin (≥1000 mg/day) monotherapy at least 4 weeks prior to Visit 1 and had failed to achieve the glucose control goal. The glucose control goal was defined as HbA1c ≤ 6.5%.
3. Male or female with child-bearing potential agreed to use an effective method of contraception approved by the investigator during the study.
4. Understood the nature of the study, and had signed informed consent form.

Exclusion criteria

1. Patients with contraindications mentioned in the Summary of Product Characteristics for vildagliptin or metformin.
2. Patients with renal dysfunction defined as creatinine clearance < 60 ml/min at Visit 1.
3. Patients with history of hepatic impairment, including but not limited to those with pretreatment AST or ALT > 3 ULN at Visit 1.
4. Female patients who needed to lactate during the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Changhua, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vildagliptin Plus Metformin (SPC)
Started | 40
Completed | 37
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics used the Intent to Treat (ITT) population: all enrolled patients who took at least one tablet of vildagliptin plus metformin 50/500 mg, and had Baseline and at least one post treatment evaluation for efficacy measurement
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: HbA1c analysis will be performed on a blood sample obtained by study personnel.
Time Frame: Baseline, Week 24
Population: Intent to Treat (ITT) population: all enrolled patients who took at least one tablet of vildagliptin plus metformin 50/500 mg, and had Baseline and at least one post treatment evaluation for efficacy measurement
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
percentage | -0.82 (0.759)

2. Secondary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c analysis will be performed on a blood sample obtained by study personnel.
Time Frame: Baseline, week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
percentage | -0.82 (0.609)

3. Secondary Outcome: Mean Change From Baseline in Fasting Plasma Glucose(FPG) at Week 12 and 24
Description: FPG analysis will be performed on a blood sample obtained by study personnel.
Time Frame: Baseline, week 12, week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
mg/dL
  Week 12 | -20.6 (25.2)
  Week 24 | -19.9 (31.9)

4. Secondary Outcome: Mean Change From Baseline in Postprandial Plasma Glucose(PPG) at Week 12 and 24
Description: PPG analysis will be performed on a blood sample obtained by study personnel.
Time Frame: Baseline, week, week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
mg/dL
  Week 12 | -40.9 (41.7)
  Week 24 | -38.3 (50.6)

5. Secondary Outcome: Mean Change From Baseline in Mean Amplitude of Glycemic Excursions (MAGE) Detected by Continuous Glucose Monitoring System (CGMS) After 24-week
Description: Mean amplitude of glycemic excursions (MAGE), which was used to quantify major swings of glycaemia and assess intra-day glycemic variability, was measured by inserting continuous glucose monitoring system (CGMS) in patients for 72 consecutive hours before Day 1 (Visit 2) and Week 24 (Visit 5). In order to unify the different initial time and time of completion in each patient, only the data recorded from Day 2 00:00 to Day 3 23:59 with total 48 hours were analyzed.
Time Frame: Baseline, week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 38
mg/dL | -12.8 (31.8)

6. Secondary Outcome: The Percentage of Patients Achieving the Two Glycemic Goals After 12- and 24-week Treatment
Description: Patients reaching glycemic goal of HbA1c ≤ 6.5% and ≤ 7.0% at week 12 and 24 will be calculated respectively.
Time Frame: week 12, week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vildagliptin Plus Metformin (SPC)
Number analyzed (Participants) | 39
percentage of participants
  HbA1c ≤ 6.5% Week 12 | 64.1
  HbA1c ≤ 6.5% Week 24 | 66.7
  HbA1c ≤ 7.0% Week 12 | 92.3
  HbA1c ≤ 7.0% Week 24 | 87.2

ADVERSE EVENTS:
Arm/Group | Vildagliptin Plus Metformin (SPC)
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin Plus Metformin (SPC) (N=40)
Pelvic cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vildagliptin Plus Metformin (SPC) (N=40)
Neutropenia (Blood and lymphatic system disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 3
Vulvovaginitis (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.